CLINICAL TRIAL: NCT04792957
Title: Expression of the JAK-STAT Signaling Pathway in Pyoderma Gangrenosum Pathological Biopsy
Brief Title: JAK-STAT Signaling Pathway in Pyoderma Gangrenosum
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ismail Sari, Professor Doctor, Dokuz Eylul University
Other Study IDs: DokuzEU-Rheumatology-1
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Pyoderma Gangrenosum; Hidradenitis Suppurativa; Psoriasis
Keywords: JAK-STAT pathway; Pyoderma Gangrenosum; Skin Biopsy
MeSH Terms: conditions — Pyoderma Gangrenosum; Hidradenitis Suppurativa; Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pyoderma Gangrenosum: Skin biopsies obtained from patients with pyoderma gangrenosum will be studied to evaluate JAK/STAT pathway by using immunohistochemical methods.
  Interventions: Diagnostic Test: immunohistochemical methods
- Hidradenitis Suppurativa: Skin biopsies obtained from patients with hidradenitis suppurativa, will be studied to evaluate JAK/STAT pathway by using immunohistochemical methods
  Interventions: Diagnostic Test: immunohistochemical methods
- Psoriasis: Skin biopsies obtained from patients with psoriasis, will be studied to evaluate JAK/STAT pathway by using immunohistochemical methods
  Interventions: Diagnostic Test: immunohistochemical methods
- Healthy Subjects: Skin biopsies obtained from patients with healthy subjects, will be used to control group.
  Interventions: Diagnostic Test: immunohistochemical methods

INTERVENTIONS:
Diagnostic Test: immunohistochemical methods — The following immunohistochemical stains will be used to evaluate the expression of JAK/STAT pathway: JAK1, JAK2, JAK3, Tyrosine Kinase 2, STAT1, STAT2, STAT3, STAT3, STAT4, STAT5 and STAT6. Staining intensity will be recorded categorically (negative and positive). The positive staining will also be graded semi-quantitively as follows: mildly positive, moderately positive and strongly positive.

SUMMARY:
The investigators hypothese that Janus kinase/signal transduction and activator of transcription (JAK/STAT) signaling pathway play a key role in pathophysiology of pyoderma gangrenosum (PG). In this study JAK/STAT signaling pathway will be investigated in the skin biopsies of PG patients

DETAILED DESCRIPTION:
Cytokines are key molecules in the pathogenesis of inflammatory diseases. These molecules exert their effects through cell surface receptors and intracellular signaling pathways. Janus kinase/signal transduction and activator of transcription (JAK/STAT) signaling pathway is implicated in the pathogenesis of several autoimmune diseases. Pyoderma gangrenosum (PG) is an inflammatory skin disease characterized by progressive and recurrent skin ulceration of destructive course. Treatment of PG requires aggressive immunosuppressive therapy but despite the use of several agents, including tumor necrosis factor inhibitory treatments there is still an unmet need in refractory PG. Recent reports suggested activation of JAK/STAT pathway in PG and some case-based studies suggested the beneficial effect of JAK-STAT inhibitory agent in the treatment of PG.

Skin biopsies obtained from PG, hidradenitis suppurativa, psoriasis and healthy subjects will be studied to evaluate JAK/STAT pathway by using immunohistochemical methods. The following immunohistochemical stains will be used to evaluate the expression of JAK/STAT pathway: JAK1, JAK2, JAK3, Tyrosine Kinase 2, STAT1, STAT2, STAT3, STAT3, STAT4, STAT5 and STAT6. Staining intensity will be recorded categorically (negative and positive). The positive staining will also be graded semi-quantitively as follows: mildly positive, moderately positive and strongly positive.

ELIGIBILITY:
Inclusion Criteria:

* Pyoderma gangrenosum diagnosed with skin biopsy
* Psoriasis diagnosed with skin biopsy
* Hidradenitis suppurativa diagnosed with skin biopsy
* Skin biopsy in healthy subjects

Exclusion Criteria:

- This is a case-based study and there is no exclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from İzmir Katip Çelebi University, Ataturk Education and Research Hospital Department of Rheumatology
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Expression of JAK-STAT pathway | 15 years
  Expression of JAK1, JAK2, JAK3, Tyrosine Kinase 2, STAT1, STAT2, STAT3, STAT3, STAT4, STAT5 and STAT6 in tissue levels in PG.